CLINICAL TRIAL: NCT03250689
Title: Randomized Double Blind (Sponsor Unblind) Study Evaluating the Effect of 14 Days of Treatment With Danirixin (GSK1325756) on Neutrophil Extracellular Traps (NETs) Formation in Participants With Stable Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Randomized Study Evaluating the Effect of Danirixin on Neutrophil Extracellular Traps (NETs) in Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to a change in the benefit-risk profile for danirixin in COPD.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207551; 2017-001069-25 (EudraCT Number)
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Results first posted 2019-11-08 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Danirixin; CXCR2; NETs; GSK1325756; COPD; HBr
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — danirixin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Danirixin 35 mg (Experimental): Eligible subjects will receive danirixin 35 mg tablet with food twice daily for 14 Days.
  Interventions: Drug: Danirixin; Drug: Rescue medication; Drug: Inhaled COPD maintenance medication
- Placebo Comparator (Experimental): Eligible subjects will receive placebo tablet with food twice daily for 14 Days.
  Interventions: Drug: Placebo; Drug: Rescue medication; Drug: Inhaled COPD maintenance medication

INTERVENTIONS:
Drug: Danirixin — Danirixin will be available as 35 mg oval shaped, white film coated HBr embossed tablets.
  Arms: Danirixin 35 mg
Drug: Placebo — Placebo will be available as oval shaped, white film coated tablets.
  Arms: Placebo Comparator
Drug: Rescue medication — Subjects may continue to use rescue medication(s) anytime during the study. The following rescue medications may be used: short acting beta agonists, short acting muscarinic antagonists, or short acting combination bronchodilators.
Drug: Inhaled COPD maintenance medication — Subjects may continue to use inhaled COPD maintenance medication(s) during the study, at the discretion of the GSK Medical Monitor and/or Investigator. The following maintenance medications may be used: long acting bronchodilator medications (e.g. long-acting muscarinic antagonist [LAMA], long-acting beta-agonist [LABA]) and long-acting bronchodilator combination therapies (e.g. LAMA/LABA) and long-acting bronchodilator/inhaled corticosteroid steroid combination (ICS) therapies (e.g. LABA/ICS, LAMA/LABA/ICS)

SUMMARY:
The inflammation associated with COPD is characterized by a prominent infiltration of neutrophils in lung tissue and airways. The CXC chemokine receptor type 2 (CXCR2) plays a pivotal role in neutrophil recruitment to the lungs resulting in progressive fibrosis, airway stenosis, and destruction of the lung parenchyma characteristic of COPD. There is a paucity of novel therapies that target these symptoms, and there are no currently available therapies that modify disease progression in COPD. Danirixin (GSK1325756) is a selective CXCR2 antagonist being developed as a potential anti-inflammatory agent for the treatment of COPD and influenza. This study is a mechanistic study which aims to evaluate the effect of danirixin in reducing neutrophil extracellular traps (NETs) formation (or NETosis). Subjects will be randomized (3:1) to receive danirixin hydrobromide (HBr) 35 milligram (mg) orally twice daily or matching placebo for 14 days. Subjects may continue to use rescue medication(s) and inhaled COPD maintenance medication(s) during the study. The study will consist of a screening period of up to 30 days, a 2 week treatment period, and a 1-week follow-up visit via phone call. Approximately 50 subjects will be screened to obtain approximately 24 subjects to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 50 to 75 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of COPD with mild to moderate airflow obstruction FEV1/FVC ratio <0.7 and FEV1% predicted (pred) >=40% at screening) based on the Quanjer reference equations, with spirometry conducted according to American Thoracic Society (ATS)/European Respiratory Society (ERS) current guidelines.
* Elevated sputum neutrophil extracellular traps based on screening assay for histone-elastase complexes of >0.5 units/ milliliter (mL) sputum. Two further screening samples can be submitted for analysis within 30 day screening period if previous samples do not pass criteria.
* Able to produce at least 1 mL of sputum sample at the screening visit with nebulized saline induction.
* Current smokers and former smokers with a cigarette smoking history of >=10 pack years (1 pack year=20 cigarettes smoked per day for 1 year or equivalent). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.
* Body weight >=45 kilogram (kg).
* Male or female.
* A male subject must agree to use contraception during the treatment period and for at least [60 hours, corresponding to approximately 6 half-lives (which is the time needed to eliminate any teratogenic treatments after the last dose of study treatment and refrain from donating sperm during this period.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and is not a woman of childbearing potential (WOCBP) OR a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 60 hours after the last dose of study treatment.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Primary clinical diagnoses of any of the following relevant lung diseases; asthma, sarcoidosis, tuberculosis, pulmonary fibrosis, severe bronchiectasis or lung cancer.
* Known alpha-1-antitrypsin deficiency.
* Pulse oximetry <88% at rest at screening. Subjects should be tested while breathing room air.
* Subjects on long term oxygen therapy (defined as >15 hours/day of oxygen use).
* Unstable co-morbidities (e.g. cardiovascular disease, active malignancy) which in the opinion of the Investigator would make the subject unsuitable to be enrolled in the study. This includes any abnormality identified on screening bloods or screening ECG which in the opinion of the Investigator would make the subject unsuitable for the study.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator of GSK medical monitor, contraindicates their participation.
* Current or chronic history of liver disease, or know hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Antibiotic use concurrently or within 28 days preceding the screening visit, including current or planned chronic use of macrolide antibiotics during the study period for the prevention of COPD exacerbations. Examples of chronic use include daily or two-three times per week for at least 3 months.
* Systemic immunosuppressive medication, including current oral corticosteroids at a dose >5 milligram (mg), concurrently or within 28 days preceding the screening visit.
* Oral or injectable Cytochrome P450 (CYP) 3A4 or Breast Cancer Resistance Protein (BCRP) substrates with narrow therapeutic index (CYP3A4 substrates include, but are not limited to, alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus, and theophylline; BCRP substrates include: Methotrexate, mitoxantrone, imatinib, irinotecan, lapatinib, rosuvastatin, sulfasalazine, topotecan.
* Current use of phosphodiesterase-4 inhibitors: Roflumilast, Crisaborole and Apremilast.
* Current use of Raloxifene.
* Current use of low molecular weight heparin.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four investigational products within 12 months prior to the first dosing day.
* Subjects with a peripheral blood neutrophil count < 1.0x10^9/liter (L) at screening.
* Diagnosis of pneumonia (chest X-ray or computed tomography [CT] confirmed) within the 3 months prior to screening.
* Chest X-ray (posterior with lateral) or CT scan reveals evidence of a clinically significant abnormality not believed to be due to the presence of COPD (historic data up to 1 year may be used).
* Abnormal and clinically significant 12-lead ECG finding at screening. The investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding that would preclude a subject from entering the trial is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following:
* AF with rapid ventricular rate > 120 beats per minute (bpm);
* Sustained or non-sustained ventricular tachycardia (VT);
* Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator has been implanted);
* QT interval corrected for heart rate by Fridericia's formula (QTcF) >=500 millisecond (msec) in subjects with QRS <120 msec and QTcF >=530 msec in subjects with QRS >=120 msec.
* Affiliation with a study site: study investigators, sub-investigators, study coordinators, employees of a study investigator, sub-investigator or study site, or immediate family members of any of the above that is involved with the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20764

REFERENCES:
- [Background] Keir HR, Richardson H, Fillmore C, Shoemark A, Lazaar AL, Miller BE, Tal-Singer R, Chalmers JD, Mohan D. CXCL-8-dependent and -independent neutrophil activation in COPD: experiences from a pilot study of the CXCR2 antagonist danirixin. ERJ Open Res. 2020 Nov 10;6(4):00583-2020. doi: 10.1183/23120541.00583-2020. eCollection 2020 Oct. PMID 33263062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in United Kingdom. This study was terminated early due to a change in the benefit risk profile of danirixin observed in another study NCT03034967, leading to cessation of the overall danirixin development program.
Pre-assignment Details: A total of 43 participants were screened, of which 23 were screen failures (23 participants did not meet inclusion/exclusion criteria). From the 20 participants who passed screening, 1 was not randomized due to study being terminated early. Hence, 19 participants were enrolled and received treatment in this study.
Groups:
- Placebo: Participants received one tablet of matching placebo twice daily orally with food for 14 days.
- Danirixin Hydrobromide 35 mg: Participants received one tablet of danirixin hydrobromide 35 milligram (mg) twice daily orally with food for 14 days.
Period: Overall Study
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Started | 5 | 14
Completed | 5 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg | Total
Number analyzed (Participants) | 5 | 14 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (6.02) | 65.3 (7.03) | 64.3 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 3 | 8 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White: White/Caucasian/European Heritage | 5 | 14 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Sputum Neutrophil Extracellular Traps (NETs) Quantified by Histone-Elastase Complexes
Description: Sputum samples were collected at indicated time points to assess NET formation via histone elastase complexes. Baseline was considered as Day 1. If Day 1 values were missing, screening value was imputed for Baseline. Change from Baseline was calculated as post-Baseline value minus Baseline value. Percentage change from Baseline was calculated by dividing change from Baseline value by Baseline value and multiplied by 100. Analysis was performed using a mixed effect repeated measures model with covariates of treatment group, log(Baseline NETs) and treatment group by day interaction. The response variable was the log of the ratio of post-Baseline NETs to Baseline NETs. Primary completer population consisted of all participants in the Modified Intent-To-Treat population who had completed the assessments supporting the primary endpoint (sputum NETs).
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: Primary Completer Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 3 | 8
Percent change
  Day 7, n=3,6: number analyzed (Participants) | 3 | 6
  Day 7, n=3,6 | -3.2 [-77.0 to 306.6] | -9.4 [-64.4 to 130.6]
  Day 14, n=3,8 | -30.5 [-71.7 to 70.7] | -13.6 [-49.1 to 46.5]

2. Secondary Outcome: Change From Baseline in Sputum NETs Quantified by Deoxyribonucleic Acid (DNA)-Elastase Complexes
Description: Sputum samples were collected at indicated time points to assess NET formation via DNA elastase complexes. Baseline was considered as Day 1. If Day 1 values were missing, screening value was imputed for Baseline. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units per milliliter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 3 | 8
Units per milliliter
  Day 7, n=3,6: number analyzed (Participants) | 3 | 6
  Day 7, n=3,6 | 1.83 (4.610) | 0.63 (1.859)
  Day 14, n=3,8 | -4.53 (2.696) | 2.08 (4.072)

3. Secondary Outcome: Change From Baseline in Percentage of Microscope Field Area Occupied by Sputum NETs
Description: Sputum samples were collected at indicated time points and NETs area was quantified by microscopy. Baseline was considered as Day 1. If Day 1 values were missing, screening value was imputed for Baseline. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: Primary Completer Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Percentage of microscope field area
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 2 | 7
Percentage of microscope field area
  Day 7 | NA (NA) — Data was not collected because 7 days treatment was insufficient to observe the changes in the sputum NETs via microscopy. | NA (NA) — Data was not collected because 7 days treatment was insufficient to observe the changes in the sputum NETs via microscopy.
  Day 14 | 0.900 (0.9200) | -0.259 (0.5183)

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes, Modified Intent-to-Treat Population consisted of all randomized participants who received at least one dose of study treatment.
Time Frame: Up to Day 21
Population: Modified Intent-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Participants
  AEs | 3 | 6
  SAEs | 0 | 0

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in seated position after 5 minutes rest for the participants at indicated time points. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Millimeters of mercury
  SBP, Day 7 | -11.2 (17.01) | -4.1 (17.70)
  SBP, Day 14 | -1.4 (16.10) | -5.3 (15.77)
  DBP, Day 7 | -2.2 (9.91) | -2.1 (10.34)
  DBP, Day 14 | 2.6 (11.01) | -5.3 (7.98)

6. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured in seated position after 5 minutes rest for the participants at indicated time points. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Beats per minute
  Day 7 | 6.8 (6.02) | 1.6 (11.28)
  Day 14 | 4.0 (6.89) | 0.1 (6.86)

7. Secondary Outcome: Change From Baseline in Respiration Rate
Description: Respiration rate was measured in seated position after 5 minutes rest for the participants at indicated time points. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Breaths per minute
  Day 7 | -0.6 (1.95) | 1.8 (2.67)
  Day 14 | 0.2 (0.84) | 2.1 (3.43)

8. Secondary Outcome: Change From Baseline in PR Interval, QRS Duration, QT Interval and QT Interval Corrected for Heart Rate According to Fridericia's Formula (QTcF)
Description: Triplicate 12-lead electrocardiograms (ECG) were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Milliseconds
  PR Interval | 7.6 (20.44) | -4.8 (15.69)
  QRS Duration | -0.3 (1.12) | 0.5 (5.55)
  QT Interval | -4.8 (10.05) | 3.7 (15.67)
  QTcF Interval | -4.6 (0.38) | -1.6 (5.96)

9. Secondary Outcome: Spirometry: Forced Expiratory Volume in One Second (FEV1) at Indicated Time Points
Description: FEV1 is the amount of air that can be forcefully exhaled from the lungs in the first second of a forced exhalation. It was measured by spirometry test. Mean and standard deviation data of FEV1 measured at Day 1 and Day 14 have been presented.
Time Frame: Day 1 and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Liter
  Day 1 | 2.458 (0.6331) | 1.914 (0.7267)
  Day 14 | 2.344 (0.7174) | 1.910 (0.7428)

10. Secondary Outcome: Spirometry: Forced Vital Capacity (FVC) at Indicated Time Points
Description: FVC is defined as the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. It was measured by spirometry test. Mean and standard deviation data of FVC measured at Day 1 and Day 14 have been presented.
Time Frame: Day 1 and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Liter
  Day 1 | 4.026 (1.2021) | 3.416 (1.1304)
  Day 14 | 4.036 (1.3992) | 3.369 (1.1456)

11. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Platelets Counts, Total Neutrophils, White Blood Cell (WBC) Count
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Platelets counts, Total neutrophils and WBC count. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Giga cells per liter
  Basophils | 0.00 (0.000) | -0.02 (0.058)
  Eosinophils | 0.040 (0.0686) | -0.020 (0.0609)
  Lymphocytes | -0.20 (0.316) | -0.08 (0.269)
  Monocytes | -0.04 (0.114) | 0.02 (0.080)
  Platelets counts | 8.2 (18.94) | -7.9 (41.66)
  Total neutrophils | -0.38 (0.965) | 0.29 (0.943)
  WBC count | -0.56 (0.948) | 0.16 (1.075)

12. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: Hematocrit. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Percentage of red blood cells in blood | -0.0058 (0.02279) | -0.0115 (0.02085)

13. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Hemoglobin. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Grams per liter | -2.2 (6.72) | -5.4 (7.99)

14. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: Mean Corpuscular Volume. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Femtoliter | 0.06 (1.339) | 0.31 (1.263)

15. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Mean Corpuscular Hemoglobin. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Picograms | -0.08 (0.920) | -0.22 (0.749)

16. Secondary Outcome: Change From Baseline in Hematology Parameter: Red Blood Cell Count
Description: Blood samples were collected to analyze the hematology parameter: Red Blood Cell count. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Trillion cells per liter | -0.070 (0.2081) | -0.154 (0.2171)

17. Secondary Outcome: Change From Baseline in Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST)
Description: Blood samples were collected to analyze the chemistry parameters: ALT, ALP and AST. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
International units per liter
  ALT | -1.6 (4.39) | -1.9 (8.24)
  ALP | 2.8 (6.26) | 1.3 (13.89)
  AST | -0.6 (2.61) | -3.1 (2.11)

18. Secondary Outcome: Change From Baseline in Chemistry Parameters: Calcium, Glucose, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameters: Calcium, Glucose, Potassium, Sodium and Urea. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Millimoles per liter
  Calcium | -0.032 (0.0782) | -0.034 (0.0947)
  Glucose | 0.36 (0.635) | 0.12 (0.398)
  Potassium | -0.12 (0.148) | 0.06 (0.287)
  Sodium | 0.0 (1.58) | 0.2 (2.04)
  Urea | -0.42 (0.867) | 0.26 (0.777)

19. Secondary Outcome: Change From Baseline in Chemistry Parameters: Creatinine, Direct Bilirubin, Total Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: Creatinine, Direct Bilirubin and Total Bilirubin. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Micromoles per liter
  Creatinine | 2.6 (5.86) | 1.2 (6.99)
  Direct Bilirubin | -0.4 (0.55) | 0.7 (1.65)
  Total Bilirubin | 0.8 (0.84) | -1.2 (3.26)

20. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urinary specific gravity measurement is a part of routine urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine. It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine samples were collected from participants at indicated time points for analysis of specific gravity. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
Unitless | 0.0030 (0.00908) | 0.0046 (0.00887)

21. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Potential of Hydrogen (pH)
Description: Urine samples were collected from participants at indicated time points for analysis of pH. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 14
pH | 1.00 (1.225) | -0.25 (0.672)

22. Secondary Outcome: Change From Baseline in Sputum Resistin Levels
Description: Sputum samples were collected at indicated time points to analyze resistin levels. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Nanograms per milliliter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 3 | 8
Nanograms per milliliter
  Day 7, n=3,6: number analyzed (Participants) | 3 | 6
  Day 7, n=3,6 | 8.93 (15.513) | -2.01 (4.629)
  Day 14, n=3,8 | 15.28 (27.619) | 2.61 (2.711)

23. Secondary Outcome: Change From Baseline in the Ratio of Sputum NETs to Sputum Neutrophils
Description: Sputum samples were collected to calculate ratio of sputum NETs to sputum neutrophils. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value. The ratio is calculated as the sputum NETs divided by the number of sputum neutrophils.
Time Frame: Baseline (Day 1) and Day 14
Population: Primary Completer Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 2 | 7
Ratio | 0.5200 (0.41000) | 0.4557 (0.53149)

24. Secondary Outcome: Change From Baseline in Sputum Elastase Activity
Description: Sputum samples were collected at indicated time points to analyze sputum elastase activity. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Nanograms per milliliter
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 3 | 8
Nanograms per milliliter
  Day 7, n=3,6: number analyzed (Participants) | 3 | 6
  Day 7, n=3,6 | 638.0 (381.36) | 238.0 (224.50)
  Day 14, n=3,8 | 411.3 (439.20) | 66.1 (45.64)

25. Secondary Outcome: Change From Baseline in Peripheral Blood Neutrophil NETs Formation Quantified by DNA Release
Description: Blood samples were collected at indicated time points to analyze peripheral blood neutrophil NETs formation by DNA release. DNA-elastase complexes quantified NETs formation. Phorbol 12-myristate 13-acetate (PMA) was used to induce inflammation and NETs formation in the PMA stimulated samples. Blood from participants were tested at Baseline and Day 14 for non-PMA stimulated samples, and at Baseline and Day 14 in PMA-stimulated samples to test whether treatment had any effect on NETs formation either naturally (non PMA induced) or where NETs formation was already raised (PMA stimulated). Hence participants were counted in both the categories - PMA stimulated and not PMA stimulated. NETs formation in peripheral blood was measured with SYTOX green fluorescence quantification of extracellular DNA. Baseline was considered as Day 1. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 14
Population: Modified Intent-to-Treat Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Relative fluorescence units
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 5 | 12
Relative fluorescence units
  Not PMA stimulated | 3044.8 (4251.78) | -721.1 (731.82)
  PMA stimulated | -96.8 (9418.43) | -1211.0 (5102.21)

26. Secondary Outcome: Percentage Change From Baseline in Peripheral Blood Neutrophil NETs Formation Quantified by Microscopy
Description: Blood samples were collected at indicated time points to analyze peripheral blood neutrophil NETs formation by microscopy.DNA-elastase complexes quantified NETs formation.PMA was used to induce inflammation and NETs formation in PMA stimulated samples. Blood from participants were tested at Baseline and Day14 for non-PMA stimulated samples,and at Baseline and Day14 in PMA-stimulated samples to test whether treatment had any effect on NETs formation either naturally(non PMA induced)or where NETs formation was already raised(PMA stimulated).Participants were counted in both categories-PMA stimulated and not PMA stimulated.NETs formation in peripheral blood was measured with SYTOX green fluorescence quantification of extracellular DNA.Baseline was considered as Day1.Change from Baseline was calculated as post-Baseline value minus Baseline value.Percentage change from Baseline was calculated by dividing change from Baseline value by Baseline value and multiplied by100.
Time Frame: Baseline (Day 1) and Day 14
Population: as for outcome 25
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 4 | 11
Percent change
  Not PMA stimulated | 927.5 (585.03) | 560.5 (395.72)
  PMA stimulated | 44.7 (41.79) | 90.6 (60.33)

27. Secondary Outcome: Maximum Observed Concentration (Cmax) of Danirixin
Description: Blood samples were collected to evaluate the pharmacokinetic (PK) of danirixin at the indicated time points for the analysis of Cmax. PK population consisted of all participants in the Modified Intent-To-Treat population who had at least 1 non-missing PK assessment (non-quantifiable values were considered as non-missing values).
Time Frame: Days 1 and 14: Pre-dose and 0.5, 1, 2 and 4 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 14
Nanograms per milliliter
  Day 1, n=14 | 855.2 (52.29)
  Day 14, n=13: number analyzed (Participants) | 13
  Day 14, n=13 | 1135.2 (65.73)

28. Secondary Outcome: Time to Cmax (Tmax) of Danirixin
Description: Blood samples were collected to evaluate the PK of danirixin at the indicated time points for the analysis of Tmax.
Time Frame: Days 1 and 14: Pre-dose and 0.5, 1, 2 and 4 hours post-dose
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours
Arm/Group | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 14
Hours
  Day 1, n=14 | 1.000 [0.50 to 4.00]
  Day 14, n=13: number analyzed (Participants) | 13
  Day 14, n=13 | 1.000 [0.50 to 4.00]

29. Secondary Outcome: Area Under the Blood Concentration-time Curve [AUC(0-t)] of Danirixin
Description: Blood samples were collected to evaluate the PK of danirixin at the indicated time points for the analysis of AUC(0-t).
Time Frame: Days 1 and 14: Pre-dose and 0.5, 1, 2 and 4 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours * nanograms per milliliter
Arm/Group | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 13
Hours * nanograms per milliliter
  Day 1 | 2173.4 (39.57)
  Day 14 | 2751.1 (51.24)

30. Secondary Outcome: Time of Last Observed Concentration (Tlast) of Danirixin
Description: Blood samples were collected to evaluate the PK of danirixin at the indicated time points for the analysis of Tlast.
Time Frame: Days 1 and 14: Pre-dose and 0.5, 1, 2 and 4 hours post-dose
Population: as for outcome 27
Measure: Median (Full Range); unit: Hours
Arm/Group | Danirixin Hydrobromide 35 mg
Number analyzed (Participants) | 14
Hours
  Day 1, n=14 | 4.000 [4.00 to 4.05]
  Day 14, n=13: number analyzed (Participants) | 13
  Day 14, n=13 | 4.000 [4.00 to 4.00]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from start of the treatment up to Day 21
Description: AEs and SAEs were collected for modified Intent-to-Treat Population which consisted of all randomized participants who received at least one dose of study treatment.
Arm/Group | Placebo | Danirixin Hydrobromide 35 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/14
Other Adverse Events (participants affected / at risk) | 3/5 | 6/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | Danirixin Hydrobromide 35 mg (N=14)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT03250689/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT03250689/SAP_001.pdf